CLINICAL TRIAL: NCT00231400
Title: Pompe Disease Registry
Brief Title: Pompe Disease Registry Protocol
Status: Recruiting | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: DIREGC07005
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Glycogen Storage Disease Type II; Pompe Disease
Keywords: Glycogen Storage Disease Type II (GSD-II); GSD-II; Pompe Disease; Pompe Disease (late-onset); Acid Maltase Deficiency Disease; Glycogenosis II
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Pompe Registry is a global, multicenter, international, longitudinal, observational, and voluntary program for patients with Pompe disease, designed to track the disease's natural history and outcomes in patients, both treated and not. Data from the Registry are also used to fulfill various global regulatory commitments, to support product development/reimbursement, and for other research and non-research related purposes.

The objectives of the Registry are:

* To enhance understanding of the variability, progression, identification, and natural history of Pompe disease, with the ultimate goal of better guiding and assessing therapeutic intervention.
* To assist the Pompe medical community with the development of recommendations for monitoring patients, and to provide reports on patient outcomes, to optimize patient care.
* To characterize the Pompe disease population.
* To evaluate the long-term effectiveness of alglucosidase alfa.

DETAILED DESCRIPTION:
Study Design Time Perspective: Retrospective and Prospective

ELIGIBILITY:
Inclusion Criteria:

All patients with a confirmed diagnosis of Pompe disease who have signed the informed consent and authorization form(s) are eligible for inclusion. Confirmed diagnosis is defined as documented GAA enzyme deficiency from blood, skin, or muscle tissue and/or documentation of 2 GAA gene mutations.

Exclusion Criteria:

There are no exclusion criteria in this Registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a confirmed diagnosis of Pompe disease are eligible for inclusion in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2004-09-15 (Actual); Primary Completion 2034-01-31 (Estimated); Study Completion 2034-01-31 (Estimated)

PRIMARY OUTCOMES:
Understanding of the variability, progression , identification and natural history of the manifestations of Pompe disease | maximum 30 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Genzyme, a Sanofi Company
Locations (272):
- United States (92):
  - University Alabama at Birmingham- Site Number : 840106, Birmingham, Alabama
  - Barrow Neurological Institute- Site Number : 840087, Phoenix, Arizona
  - Phoenix Children's Hospital- Site Number : 840003, Phoenix, Arizona
  - University of Arizona- Site Number : 840015, Tucson, Arizona
  - Arkansas Childrens Hospital- Site Number : 840109, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences- Site Number : 840113, Little Rock, Arkansas
  - University of California at Irvine- Site Number : 840036, Irvine, California
  - Loma Linda University- Genetics- Site Number : 840070, Loma Linda, California
  - Southern California Permanente Medical Group- Site Number : 840108, Los Angeles, California
  - USC Health Sciences Center Dept of Genetics- Site Number : 840082, Los Angeles, California
  - Children's Hospital Oakland- Site Number : 840029, Oakland, California
  - Children's Hospital of Orange County- Site Number : 840074, Orange, California
  - UC Davis MIND Institute- Site Number : 840010, Sacramento, California
  - University of California at San Diego- Site Number : 840007, San Diego, California
  - University of California at San Francisco- Site Number : 840051, San Francisco, California
  - Stanford University Pediatrics- Site Number : 840021, Stanford, California
  - Children's Hospital Colorado - Aurora- Site Number : 840069, Aurora, Colorado
  - Yale - Site Number : 840047, New Haven, Connecticut
  - Children's National Medical Center- Site Number : 840067, Washington D.C., District of Columbia
  - University of Florida College of Medicine- Site Number : 840012, Gainesville, Florida
  - University of Florida Pediatrics Genetics- Site Number : 840121, Jacksonville, Florida
  - University Of Miami SOM- Site Number : 840006, Miami, Florida
  - University of Florida-Genetics- Site Number : 840096, Tampa, Florida
  - Emory University School of Medicine- Human Genetics- Site Number : 840060, Decatur, Georgia
  - University of Colorado at Denver Genetics- Site Number : 840068, Aurora, Illinois
  - Ann and Robert Lurie Children's Hospital- Site Number : 840011, Chicago, Illinois
  - Ann and Robert Lurie Children's Hospital- Site Number : 840013, Chicago, Illinois
  - Rush University Medical Center Genetics- Site Number : 840079, Chicago, Illinois
  - Indianapolis University School of Medicine- Site Number : 840027, Indianapolis, Indiana
  - University of Iowa- Site Number : 840032, Iowa City, Iowa
  - University of Kansas Medical Center- Site Number : 840020, Kansas City, Kansas
  - University of Louisville- Genetics- Site Number : 840030, Louisville, Kentucky
  - Maine Medical Center Pediatrics- Site Number : 840064, Portland, Maine
  - John Hopkins- Site Number : 840044, Baltimore, Maryland
  - Massachusetts General Hospital-Genetics- Site Number : 840062, Boston, Massachusetts
  - Boston Children's Hospital - PIN- Site Number : 840092, Boston, Massachusetts
  - Baystate Health- Site Number : 840002, Springfield, Massachusetts
  - University of Michigan Pediatrics- Site Number : 840107, Ann Arbor, Michigan
  - Children's Hospital of Michigan- Site Number : 840066, Detroit, Michigan
  - Spectrum for Health- Site Number : 840019, Grand Rapids, Michigan
  - Infusion Associates- Site Number : 840050, Grand Rapids, Michigan
  - Children's Hospital and Clinics of Minnesota- Site Number : 840046, Minneapolis, Minnesota
  - Children's Hospitals and Clinics of Minnesota- Site Number : 840114, Minneapolis, Minnesota
  - University of Minnesota Medical Center Pediatrics- Site Number : 840035, Minneapolis, Minnesota
  - University of Minnesota Medical Center Pediatrics- Site Number : 840076, Minneapolis, Minnesota
  - University of Missouri Health System Department of Genetics- Site Number : 840031, Columbia, Missouri
  - Children's Mercy Hospital- Pediatrics- Site Number : 840063, Kansas City, Missouri
  - Washington University of St. Louis- Site Number : 840100, St Louis, Missouri
  - University of Nebraska Medical Center- Pediatrics- Site Number : 840084, Omaha, Nebraska
  - Children's Specialty Center of Nevada- Site Number : 840008, Las Vegas, Nevada
  - Cooper Health Center- Site Number : 840098, Camden, New Jersey
  - Hackensack University Medical Center- Site Number : 840101, Hackensack, New Jersey
  - Atlantic Health System- Site Number : 840099, Morristown, New Jersey
  - St. Peter's University Hospital- Site Number : 840016, New Brunswick, New Jersey
  - St. Joseph's Children's Hospital- Site Number : 840057, Paterson, New Jersey
  - Northwell Health- Site Number : 840102, Manhasset, New York
  - New York University School Of Medicine- Site Number : 840040, New York, New York
  - Metropolitan Hospital Center- Site Number : 840110, New York, New York
  - Mt. Sinai School of Medicine- Site Number : 840005, New York, New York
  - University of Rochester Medical Center SOM- Site Number : 840105, Rochester, New York
  - State University of New York- Site Number : 840052, Syracuse, New York
  - New York Medical College- Site Number : 840039, Valhalla, New York
  - Carolinas Medical Center Hospital- Site Number : 840065, Charlotte, North Carolina
  - Duke University Medical Center Genetics Dept- Site Number : 840037, Durham, North Carolina
  - University of Cincinnati Medical Center- Site Number : 840124, Cincinnati, Ohio
  - Cincinnati Children's Hospital-Genetics- Site Number : 840041, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center- Site Number : 840119, Cleveland, Ohio
  - Cleveland Clinic Foundation Pediatrics- Site Number : 840048, Cleveland, Ohio
  - Nationwide Children's Hospital - PIN- Site Number : 840091, Columbus, Ohio
  - LSD Data Registry Site LLC- Site Number : 840094, Dublin, Ohio
  - Oregon Health & Sciences University- Site Number : 840080, Portland, Oregon
  - Oregon Health & Science University (OHSU)- Site Number : 840095, Portland, Oregon
  - Oregon Health and Scinece University- Site Number : 840038, Portland, Oregon
  - Penn Hershey Medical Center- Site Number : 840061, Hershey, Pennsylvania
  - Penn State Health Milton South Hershey Medical Center- Site Number : 840126, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia HUP Medical Genetics- Site Number : 840089, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia- Site Number : 840034, Philadelphia, Pennsylvania
  - UPMC- Site Number : 840014, Pittsburgh, Pennsylvania
  - University of Pittsburgh- Site Number : 840023, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Genetics- Site Number : 840053, Providence, Rhode Island
  - Greenwood Genetcs- Site Number : 840055, Greenville, South Carolina
  - Vanderbilt University Hospital-Pediatrics- Site Number : 840049, Nashville, Tennessee
  - Baylor Research Center- Site Number : 840058, Dallas, Texas
  - Cook Children's Health Care System- Site Number : 840024, Fort Worth, Texas
  - University of Utah Department of Medical Genetics- Site Number : 840043, Salt Lake City, Utah
  - University of Virginia School of Medicine-Pediatrics- Site Number : 840078, Charlottesville, Virginia
  - O&O Alpan, LLC- Site Number : 840025, Fairfax, Virginia
  - Children's Hospital of the Kings Daughters- Site Number : 840072, Norfolk, Virginia
  - Seattle Children's Hospital- Site Number : 840028, Seattle, Washington
  - University Of Washington Medical Center- Site Number : 840059, Seattle, Washington
  - Multicare Health System ¿ Mary Bridge Childrens Hospital- Site Number : 840115, Tacoma, Washington
  - Children's Hospital of Wisconsin-Pediatrics- Site Number : 840054, Milwaukee, Wisconsin
- Argentina (4):
  - Investigational Site Number : 153195, Caba, Buenos Aires, Buenos Aires
  - Investigational Site Number : 152218, CABA, Buenos Aires
  - Investigational Site Number : 153194, CABA, Buenos Aires
  - Investigational Site Number : 153032, Ciudad Autónoma de Buenos Aires, Buenos Aires
- Australia (5):
  - Investigational Site Number : 036013, Westmead, New South Wales
  - Investigational Site Number : 151069, Westmead, New South Wales
  - Investigational Site Number : 154087, Brisbane, Queensland
  - Investigational Site Number : 152096, Brisbane, Queensland
  - Investigational Site Number : 151015, Murdoch, Western Australia
- Belgium (9):
  - Investigational Site Number : 150722, Antwerp
  - Investigational Site Number : 154298, Bruges
  - Investigational Site Number : 150684, Brussels
  - Investigational Site Number : 056010, Brussels
  - Investigational Site Number : 152072, Edegem
  - Investigational Site Number : 152295, Ghent
  - Investigational Site Number : 153179, Gosselies
  - Investigational Site Number : 151668, Leuven
  - Investigational Site Number : 152126, Leuven
- Brazil (8):
  - Hospital Universitario Walter Cantidio- Site Number : 076011, Fortaleza, Ceará
  - Hospital Geral e Maternidade de Cuiabá- Site Number : 076003, Cuiabá, Mato Grosso
  - Hospital de Clinicas de Porto Alegre- Site Number : 076008, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto- Site Number : 076009, Ribeirão Preto, São Paulo
  - Instituto Fernandes Figueira - FIOCRUZ- Site Number : 076001, Rio de Janeiro
  - Instituto de Genética e Erros Inatos do Metabolismo- Site Number : 076002, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo- Site Number : 076004, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo- Site Number : 076007, São Paulo
- Investigational Site Number : 100001, Sofia, Bulgaria
- Canada (12):
  - Investigational Site Number : 124014, Calgary, Alberta
  - Investigational Site Number : 124002, Edmonton, Alberta
  - Investigational Site Number : 124010, Vancouver, British Columbia
  - Investigational Site Number : 124011, Vancouver, British Columbia
  - Investigational Site Number : 124019, Winnipeg, Manitoba
  - Investigational Site Number : 124022, Moncton, New Brunswick
  - Investigational Site Number : 124007, Hamilton, Ontario
  - Investigational Site Number : 124021, London, Ontario
  - Investigational Site Number : 124006, Toronto, Ontario
  - Investigational Site Number : 124004, Montreal, Quebec
  - Investigational Site Number : 124018, Montreal, Quebec
  - Investigational Site Number : 124001, Sherbrooke, Quebec
- Chile (2):
  - Investigational Site Number : 152002, Punta Arenas
  - Investigational Site Number : 152001, Santiago
- China (8):
  - Investigational Site Number : 152380, Beijing
  - Investigational Site Number : 153202, Beijing
  - Investigational Site Number : 153203, Beijing
  - Investigational Site Number : 152379, Guangzhou
  - Investigational Site Number : 152381, Jinan
  - Investigational Site Number : 157250, Jinan
  - Investigational Site Number : 152356, Shanghai
  - Investigational Site Number : 152382, Shanghai
- Investigational Site Number : 170001, Bogotá, Colombia
- Croatia (2):
  - Investigational Site Number : 1910001, Zagreb
  - Investigational Site Number : 1910002, Zagreb
- Investigational Site Number : 150809, Prague, Czechia
- Investigational Site Number : 151229, København Ø, Denmark
- France (19):
  - Investigational Site Number : 250010, Bordeaux
  - Investigational Site Number : 250012, Brest
  - Investigational Site Number : 250003, Bron
  - Investigational Site Number : 250007, Bron
  - Investigational Site Number : 250009, Caen
  - Investigational Site Number : 250015, La Tronche
  - Investigational Site Number : 250008, Lille
  - Investigational Site Number : 250002, Marseille
  - Investigational Site Number : 250017, Nancy
  - Investigational Site Number : 250019, Nantes
  - Investigational Site Number : 250005, Nice
  - Investigational Site Number : 250011, Nîmes
  - Investigational Site Number : 250004, Paris
  - Investigational Site Number : 250001, Paris
  - Investigational Site Number : 250018, Saint-Priest-en-Jarez
  - Investigational Site Number : 250016, Strasbourg
  - Investigational Site Number : 250014, Toulouse
  - Investigational Site Number : 250006, Tours
  - Investigational Site Number : 25013, Vannes
- Germany (12):
  - Investigational Site Number : 152041, Berlin
  - Investigational Site Number : 151686, Berlin
  - Investigational Site Number : 152293, Berlin
  - Investigational Site Number : 152234, Bochum
  - Investigational Site Number : 152200, Bonn
  - Investigational Site Number : 152108, Freiburg im Breisgau
  - Investigational Site Number : 154150, Giessen
  - Investigational Site Number : 152045, Halle
  - Investigational Site Number : 154215, Hamburg
  - Investigational Site Number : 150031, Mainz
  - Investigational Site Number : 152075, München
  - Investigational Site Number : 152299, Münster
- Investigational Site Number : 300001, Thessaloniki, Greece
- Investigational Site Number : 344001, Kowloon, Hong Kong
- Hungary (3):
  - Investigational Site Number : 3480009, Debrecen
  - Investigational Site Number : 3480007, Nyíregyháza
  - Investigational Site Number : 3480011, Pécs
- India (4):
  - Investigational Site Number : 356003, Ahmedabad
  - Investigational Site Number : 356001, Kolkata
  - Investigational Site Number : 3560004, Secunderabad
  - Investigational Site Number : 356002, Vellore
- Investigational Site Number : 360001, Jakarta, Indonesia
- Israel (3):
  - Investigational Site Number : 3760002, Beersheba
  - Investigational Site Number : 3760001, Haifa
  - Investigational Site Number : 3760003, Tel Aviv
- Italy (19):
  - Investigational Site Number : 380007, Milan, Milano
  - Investigational Site Number : 380011, Padua, Padova
  - Investigational Site Number : 380008, Brescia
  - Investigational Site Number : 380006, Cagliari
  - Investigational Site Number : 380014, Ferrara
  - Investigational Site Number : 380005, Florence
  - Investigational Site Number : 380004, Genova
  - Investigational Site Number : 380013, Messina
  - Investigational Site Number : 380016, Milan
  - Investigational Site Number : 380009, Monza
  - Investigational Site Number : 380010, Napoli
  - Investigational Site Number : 380019, Napoli
  - Investigational Site Number : 380002, Padua
  - Investigational Site Number : 380003, Pavia
  - Investigational Site Number : 157218, Pisa
  - Investigational Site Number : 380015, Roma
  - Investigational Site Number : 380012, Roma
  - Investigational Site Number : 380017, Torino
  - Investigational Site Number : 380001, Udine
- Japan (2):
  - Investigational Site Number : 392106, Sakyo-ku, Kyoto
  - Investigational Site Number : 392105, Ginowan, Okinawa
- Investigational Site Number : 4000001, Amman, Jordan
- Investigational Site Number : 154225, Kuwait City, Kuwait
- Investigational Site Number : 4220004, Beirut, Lebanon
- Malaysia (2):
  - Investigational Site Number : 458002, Kuala Lumpur
  - Investigational Site Number : 458001, Kuala Pahang
- Investigational Site Number : 152029, Rotterdam, Netherlands
- Pakistan (2):
  - Investigational Site Number : 154264, Karachi
  - Investigational Site Number : 154266, Lahore
- Investigational Site Number : 608001, Manila, Philippines
- Investigational Site Number : 150575, Warsaw, Poland
- Portugal (2):
  - Investigational Site Number : 620008, Coimbra
  - Investigational Site Number : 620006, Lisbon
- Investigational Site Number : 154099, Bucharest, Romania
- Investigational Site Number : 643002, Moscow, Russia
- Saudi Arabia (2):
  - Investigational Site Number : 682001, Al Qaţīf
  - Investigational Site Number : 682004, Mecca
- Investigational Site Number : 6880001, Belgrade, Serbia
- Investigational Site Number : 702001, Singapore, Singapore
- Investigational Site Number : 703001, Bratislava, Slovakia
- South Korea (9):
  - Investigational Site Number : 153178, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 153180, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 153196, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 153176, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 153191, Daejeon
  - Investigational Site Number : 153192, Seoul
  - Investigational Site Number : 151149, Seoul
  - Investigational Site Number : 153212, Seoul
  - Investigational Site Number : 153222, Seoul
- Taiwan (14):
  - Investigational Site Number : 151500, Chiayi City
  - Investigational Site Number : 154093, Chiayi City
  - Investigational Site Number : 152152, Hualien City
  - Investigational Site Number : 152244, Kaohsiung City
  - Investigational Site Number : 152246, Kaohsiung City
  - Investigational Site Number : 151534, New Taipei City
  - Investigational Site Number : 151181, Taichung
  - Investigational Site Number : 151179, Taichung
  - Investigational Site Number : 153248, Tainan
  - Investigational Site Number : 152153, Tainan
  - Investigational Site Number : 151182, Taipei
  - Investigational Site Number : 152321, Taipei
  - Investigational Site Number : 152226, Taipei
  - Investigational Site Number : 153158, Tao Yuan County
- Thailand (5):
  - Investigational Site Number : 764002, Bangkok
  - Investigational Site Number : 764003, Bangkok
  - Investigational Site Number : 764004, Bangkok
  - Investigational Site Number : 764001, Bangkok
  - Investigational Site Number : 764005, Khon Kaen
- Investigational Site Number : 7840001, Dubai, United Arab Emirates
- United Kingdom (11):
  - Investigational Site Number : 151340, Cambridge, Cambridgeshire
  - Investigational Site Number : 152334, Cardiff, Cardiff [Caerdydd Gb-crd]
  - Investigational Site Number : 150964, Salford, Manchester
  - Investigational Site Number : 152287, Birmingham
  - Investigational Site Number : 154240, Birmingham
  - Investigational Site Number : 152156, Glasgow
  - Investigational Site Number : 151123, London
  - Investigational Site Number : 151646, London
  - Investigational Site Number : 150303, London
  - Investigational Site Number : 150455, Manchester
  - Investigational Site Number : 152087, Newcastle
- Vietnam (2):
  - Investigational Site Number : 154212, Hanoi
  - Investigational Site Number : 704002, Ho Chi Minh City

REFERENCES:
- [Background] Kishnani PS, Amartino HM, Lindberg C, Miller TM, Wilson A, Keutzer J. Methods of diagnosis of patients with Pompe disease: Data from the Pompe Registry. Mol Genet Metab. 2014 Sep-Oct;113(1-2):84-91. doi: 10.1016/j.ymgme.2014.07.014. Epub 2014 Jul 16. PMID 25085280
- [Background] Kishnani PS, Amartino HM, Lindberg C, Miller TM, Wilson A, Keutzer J; Pompe Registry Boards of Advisors. Timing of diagnosis of patients with Pompe disease: data from the Pompe registry. Am J Med Genet A. 2013 Oct;161A(10):2431-43. doi: 10.1002/ajmg.a.36110. Epub 2013 Aug 30. PMID 23997011
- [Background] Byrne BJ, Kishnani PS, Case LE, Merlini L, Muller-Felber W, Prasad S, van der Ploeg A. Pompe disease: design, methodology, and early findings from the Pompe Registry. Mol Genet Metab. 2011 May;103(1):1-11. doi: 10.1016/j.ymgme.2011.02.004. Epub 2011 Feb 11. PMID 21439876
- [Derived] Berger KI, Chien YH, Dubrovsky A, Kishnani PS, Llerena JC Jr, Neilan E, Roberts M, Sheng B, Batista JL, Periquet M, Wilson KM, van der Ploeg AT. Changes in forced vital capacity over </= 13 years among patients with late-onset Pompe disease treated with alglucosidase alfa: new modeling of real-world data from the Pompe Registry. J Neurol. 2024 Aug;271(8):5433-5446. doi: 10.1007/s00415-024-12489-9. Epub 2024 Jun 19. Erratum In: J Neurol. 2025 Jul 31;272(8):547. doi: 10.1007/s00415-025-13147-4. PMID 38896264
- [Derived] Zhao Y, Wang Z, Lu J, Gu X, Huang Y, Qiu Z, Wei Y, Yan C. Characteristics of Pompe disease in China: a report from the Pompe registry. Orphanet J Rare Dis. 2019 Apr 3;14(1):78. doi: 10.1186/s13023-019-1054-0. PMID 30943998